CLINICAL TRIAL: NCT01042782
Title: Phase I Study of Daily RAD001 Administered Orally in Combination With Mitomycin C, Administered Every Three Weeks to Patients With Advanced Gastric Cancer or Cancer of the Esophagogastric Junction
Brief Title: Phase I Study of Daily RAD001 in Combination With Mitomycin C in Patients With Advanced Gastric Cancer or Cancer of the Esophagogastric Junction
Acronym: S387
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Krankenhaus Nordwest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001C24126
Record Dates: First submitted 2010-01-05; First posted 2010-01-06 (Estimated); Last update posted 2012-08-03 (Estimated); Status verified 2012-08

CONDITIONS: Advanced Gastric Cancer; Advanced Cancer of the Esophagogastric Junction
Keywords: gastric cancer; RAD001; Mitomycin C; MTD
MeSH Terms: conditions — Stomach Neoplasms | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RAD-MitC (Experimental): RAD001 orally daily 5mg or 7.5mg or 10mg Mitomycin C 5mg/m2 every 3 weeks
  Interventions: Drug: RAD001 and MitomycinC

INTERVENTIONS:
Drug: RAD001 and MitomycinC — RAD001 tablets daily, 5mg, 7.5 mg or 10 mg (3 cohorts)
  Mitomycin C 5 mg/m2 i.v. every 3 weeks
  Other Names: RAD001 (everolimus)

SUMMARY:
Patients with advanced gastric cancer are treated with a combination of RAD001 (everolimus) and Mitomycin C.

DETAILED DESCRIPTION:
The purpose of this monocenter, single-arm, phase I trial is to determine the maximum-tolerated-dose, dose-limiting toxicity (DLT) and preliminary efficacy and safety of RAD001 in combination with Mitomycin C in patients with advanced gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1 prior platin containing chemotherapy in the palliativ setting or progressive disease under adjuvant or neoadjuvant therapy within 6 months of treatment start date.
* Histological evidence of advanced or metastatic gastric cancer or cancer of the esophageal junction.
* At baseline CT or MRI scan must demonstrate measurable disease by RECIST criteria, i.e., the presence of at least one measurable lesion. Measurable disease lesions must be accurately measured in at least one dimension with longest diameter > 20 mm using conventional techniques or > 10 mm with spiral CT scan (with minimum lesion size no less than double the slice thickness).
* At least one measurable lesion outside of the field of any prior radiation therapy (according to RECIST criteria). Prior radiotherapy to a single index lesion is not allowed.
* Adult male or female patients (≥18 years of age).
* Patients must have disease not amenable to surgery, radiation, or combined modality therapy with curative intent.
* ECOG 0 or 1
* Life expectance >4 months
* Adequate bone marrow function, renal function, liver function
* Women using an acceptable form of contraception prior to receiving RAD001 or women who meet the protocol definition of post-menopausal: 12 months of natural (spontaneous) amenorrhea or 6 months of spontaneous amenorrhea with serum FSH levels >40 mIU/m or 6 weeks post surgical bilateral oophorectomy with or without hysterectomy.
* Fully recovered from any previous surgery, prior chemotherapy or radiation therapy (at least 4 weeks since major surgery or prior myelosuppressive chemotherapy). With the exception of alopecia, patients must have resolution of all acute toxic effects of any prior surgery, radiotherapy, or chemotherapy to NCI CTC (Version 2.0) grade <=1. Patients with rapidly progressive tumors (upon the decision of the investigator) can be treated <4 weeks since last chemotherapy, if they fully recovered from all side effects.
* Signed informed consent

Exclusion Criteria:

* Anticancer therapy within 3 weeks of enrollment including chemotherapy, hormonal therapy, immunotherapy, or radiotherapy. Patients with rapidly progressive tumors (upon the decision of the investigator) can be treated <4 weeks since last chemotherapy, if they fully recovered from all side effects.
* Prior therapy with RAD001 (everolimus) or other rapamycins (sirolimus, temsirolimus).
* Patients treated with Mitomycin C
* No neurotoxicity >= grade 2 CTC
* No gastric or intestinal obstruction
* Patients taking drugs known to inhibit or induce isoenzyme CYP3A
* Patients with any concurrent major medical condition liable to compromise the patient's participation in the study (e.g known HIV infection, uncontrolled diabetes, serious cardiac dysrhythmia or condition, New York Heart Association classification of III or IV, congestive cardiac failure, myocardial infarction within 6 months, unstable angina, chronic or acute renal or liver disease, uncontrolled serious infections including abscess or fistulae, etc.)
* Patients with a history of another malignancy prior to study entry, except curatively treated non-melanotic skin cancer or carcinoma in-situ cervical cancer unless in complete remission or no evidence of disease and off all therapy for that disease for a minimum of 5 years
* No symptomatic brain metastasis.
* Use of other investigational drugs at the time of enrollment, or within 30 days or 5 half-lives of enrollment, whichever is longer.
* Female patients who are pregnant or breast feeding
* History of hypersensitivity to any of the study drugs or to drugs with similar chemical structures
* History of malignancy of any organ system, treated or untreated, within the past 5 years whether or not there is evidence of local recurrence or metastases, with the exception of localized basal cell carcinoma of the skin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2008-01; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
maximum tolerated-dose (MTD) of RAD001 in combination with Mitomycin C | every week

SECONDARY OUTCOMES:
preliminary efficacy of RAD001 in refractory gastric cancer. Efficacy is defined as complete response or partial response at 12 weeks based on RECIST-criteria | every 6 weeks
progression-free survival (PFS) | every 6 weeks
overall survival (OS) | every three months
safety and tolerability of the combination of RAD001 and Mitomycin C as assessed by frequency, severity, and duration of treatment-related adverse effects | every week

CONTACTS AND LOCATIONS:
Overall Officials: Salah-Eddin Al-Batran, MD, Principal Investigator — Krankenhaus Nordwest
Locations (1):
- Krankenhaus Nordwest, Frankfurt, Germany

REFERENCES:
- [Derived] Werner D, Atmaca A, Pauligk C, Pustowka A, Jager E, Al-Batran SE. Phase I study of everolimus and mitomycin C for patients with metastatic esophagogastric adenocarcinoma. Cancer Med. 2013 Jun;2(3):325-33. doi: 10.1002/cam4.77. Epub 2013 Apr 2. PMID 23930209